CLINICAL TRIAL: NCT02097576
Title: Effectiveness of Manuka Honey/Saline Nasal Rinses as an Adjunct to Standard Medical Therapy for Chronic Rhinosinusitis: A Prospective Clinical Trial
Brief Title: Manuka Honey Nasal Rinse Study
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding withdrawn.
Sponsor: University of Florida (Other)
Collaborators: NeilMed Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014Leon
Record Dates: First submitted 2014-03-24; First posted 2014-03-27 (Estimated); Last update posted 2020-04-27 (Actual); Status verified 2020-04

CONDITIONS: Rhinosinusitis
Keywords: Chronic Rhinosinusitis
MeSH Terms: conditions — Rhinosinusitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- NeilMed Saline Sinus Rinse (Active Comparator): Saline nasal rinses will be performed using a NeilMed® Sinus Rinse 240 ml bottle and one NeilMed® packet containing sodium chloride/sodium bicarbonate at a concentration to make an isotonic solution when mixed with distilled or previously boiled water.
  Interventions: Other: NeilMed Saline Sinus Rinse
- Saline mixed with Manuka Honey (Active Comparator): Saline mixed with MH nasal rinses participants will be instructed how to mix a rounded teaspoon of MH (Wedderspoon® 100% Raw Manuka Honey Active 16+) with 4-6 oz of lukewarm distilled or previously boiled water, to add along with distilled or previously boiled water and the NeilMed® Sinus Rinse packet to the rinse bottle to a final volume of 240 ml. Participants will be instructed to rinse slowly with the MH/saline rinse mixture to maximize contact time with the MH/saline mixture.
  Interventions: Other: Saline mixed with Manuka Honey

INTERVENTIONS:
Other: Saline mixed with Manuka Honey — Saline mixed with MH nasal rinses participants will be instructed how to mix a rounded teaspoon of MH (Wedderspoon® 100% Raw Manuka Honey Active 16+) with 4-6 oz of lukewarm distilled or previously boiled water, to add along with distilled or previously boiled water and the NeilMed® Sinus Rinse packet to the rinse bottle to a final volume of 240 ml. Participants will be instructed to rinse slowly with the MH/saline rinse mixture to maximize contact time with the MH/saline mixture.
  Other Names: NeilMed® Sinus Rinse; Manuka Honey
  Arms: Saline mixed with Manuka Honey
Other: NeilMed Saline Sinus Rinse — Saline nasal rinses will be performed using a NeilMed® Sinus Rinse 240 ml bottle and one NeilMed® packet containing sodium chloride/sodium bicarbonate at a concentration to make an isotonic solution when mixed with distilled or previously boiled water.
  Arms: NeilMed Saline Sinus Rinse

SUMMARY:
The purpose of this study is to evaluate whether high-volume nasal rinses with a manuka honey/saline mixture will improve symptom scores, nasal endoscopic findings and CT scan findings compared to nasal saline rinse without manuka honey in patients with chronic rhinosinusitis.

Manuka honey is a honey made from bees that drink the nectar from tea (manuka) trees in New Zealand. It has been shown to have antibacterial activity against common bacteria that cause chronic sinusitis.

DETAILED DESCRIPTION:
If the subject chooses to participate in the study, the subject will be asked to fill out a symptom questionnaire at the beginning of the study and at each follow-up visit. The subject will be randomly assigned (much like the flip of a coin) to one of two treatment arms in addition to the prescribed medical treatments: 1) nasal rinses twice daily with a saline solution (standard therapy) or 2) nasal rinses with a saline solution mixed with manuka honey (the experimental therapy.) Subjects in the manuka honey/saline rinse arm will perform the experimental rinses twice daily for one month, and then will continue with saline rinses twice daily, with manuka honey added to the rinses only as needed. Nasal rinsing of some kind will be continued through the entire study period.

ELIGIBILITY:
Inclusion Criteria:

* Chronic Rhinosinusitis
* Nasal Polyposis stages 1-3

Exclusion Criteria:

* Nasal Polyposis stage 4-5
* Cystic Fibrosis
* Immunocompromised patients
* Allergy to bees or honey

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-05; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Change in SNOT-22 Symptomatic Scores at 1 month | Change from baseline at 1 month
  There are 22 questions, each scored 0 - 5. Possible scores are 0 - 110. The best score is 0, the worst score is 110.
Change in SNOT-22 Symptomatic Scores at 3 months | Change from baseline at 3 months
  There are 22 questions, each scored 0 - 5. Possible scores are 0 - 110. The best score is 0, the worst score is 110.
Change in SNOT-22 Symptomatic Scores at 6 months | Change from baseline at 6 months
  There are 22 questions, each scored 0 - 5. Possible scores are 0 - 110. The best score is 0, the worst score is 110.

SECONDARY OUTCOMES:
Change in Endoscopic Scores of CRS severity in the different treatment arms at 1 month | Change in baseline at 1 month
Change in Endoscopic Scores of CRS severity in the different treatment arms at 3 months | Change in baseline at 3 months
Change in Endoscopic Scores of CRS severity in the different treatment arms at 6 months | Change in baseline at 6 months
Change in Radiologic Scores of CRS severity in the different treatment arms at 3 months | Change in baseline at 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Leon, MD, Principal Investigator — University of Florida, Department of Otolaryngology; Elizabeth Leon, MD, Principal Investigator — Malcom Randall VA Medical Center